CLINICAL TRIAL: NCT06444308
Title: Assessing the Efficacy and Safety of Community Health Worker-led Hypertension Management Enabled by a Mobile Clinical Decision Support Application Compared to Physician Care: a Randomized, Controlled, Noninferiority Trial
Brief Title: Community Health Worker-led Hypertension Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0566; A532050 (Other: UW Madison); Protocol Version 1/12/26 (Other: UW Madison); 4R33TW011891-03 (NIH)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: community health worker
MeSH Terms: conditions — Hypertension | interventions — Compact Disks

STUDY DESIGN:
Intervention Model Description: cluster randomized, controlled, non-inferiority trial, each of 15 clusters of geographically grouped communities in the San Lucas Toliman municipality of Guatemala will be randomized to either CHW or physician care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker Care (Experimental): Multimodal health systems intervention: hypertension management by trained CHWs equipped with a mobile clinical decision support (CDS) application and remote supervision and support by physicians. CHWs will meet with patients each month and, with the assistance of the CDS application, follow physician-approved and evidence-based protocols to initiate and titrate antihypertensives and medications to reduce cardiovascular risk; identify potential complications of hypertension or problems with medications; and provide lifestyle counseling. For patients with comorbid hypertension and diabetes, CHWs will also manage glycemic therapy and assess for diabetes complications with the assistance of the application.
  Interventions: Other: CommCare with Mobile Clinical Decision Support (CDS) Application; Other: Remote Supervision by Physicians
- Physician Care (Active Comparator)
  Interventions: Other: CommCare Application without CDS

INTERVENTIONS:
Other: CommCare with Mobile Clinical Decision Support (CDS) Application — For those assigned to the CHW arm, management will be assisted by CDS from the CommCare application.
  Arms: Community Health Worker Care
Other: Remote Supervision by Physicians — teleconsultation with a supervising physician
  Arms: Community Health Worker Care
Other: CommCare Application without CDS — The physician will have received training and orientation on the same clinical protocols followed by the CHWs, as well as access to reference materials for these protocols, but the version of the CommCare application used will not provide CDS, but will serve to record and review patient data only.
  Arms: Physician Care

SUMMARY:
This study is to determine if hypertension management by community health workers (CHW) supported by a mobile health application and remote physician supervision is non-inferior to management by a physician for the primary outcome of improvement in systolic blood pressure. The target population is patients with hypertension in rural Guatemala. Study duration will be 12-24 months.

DETAILED DESCRIPTION:
The investigators have developed an innovative system of care utilizing CHWs equipped with a mobile application and supported and supervised remotely by physicians. This model of care is adapted from a CHW-led diabetes program enabled by a similar CDS application which the investigators implemented in the same communities in rural Guatemala where we will carry out this proposed study. This program safely led to significant improvements in glycemic control. The mobile application is built on the widely-used CommCare platform and provides clinical decision support (CDS) to CHWs based on protocols from the WHO and the International Society of Hypertension for antihypertensive medication initiation and titration, lifestyle counseling, and identification of patients requiring a higher level of care.

The Primary Objective is to determine if hypertension management by CHWs is non-inferior to care provided directly by a physician.

The Secondary Objective is to evaluate the safety, acceptability to patients, and cost of CHW-led care compared to care provided directly by a physician.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or greater with diagnosis of hypertension AND blood pressure (BP) greater than or equal to 140/90 OR currently taking antihypertensive medication.
* Ability to provide informed consent

Exclusion Criteria:

* Pregnancy
* Severe comorbid condition(s) with life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)

SECONDARY OUTCOMES:
Proportion of Participants with SBP less than 140mmHg | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Proportion of Participants with SBP less than their personalized goal | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in Diastolic Blood Pressure (DBP) | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in Hemoglobin A1c (HbA1c) | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in Diabetes Control | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  Indicated by the proportion of diabetic patients with HbA1c less than 8 and the proportion of diabetic patients with HbA1c less than their personalized goal.
Change in Weight | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in Total Cholesterol | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in LDL Cholesterol | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in HDL Cholesterol | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in Triglycerides | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in Creatinine | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in Estimated Glomerular Filtration Rate (eGFR) | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in 10 year CVD risk (per WHO risk prediction charts) | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
Change in Hypertension Self-Care Activity Level Effects (H-SCALE): Medication Adherence Subscale Score | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  The H-SCALE: Medication Adherence subscale is scored from 0-21 where higher scores indicate a more positive attitude toward adherence.
Change in H-SCALE: Weight Management Score | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  The H-SCALE: Weight Management subscale is scored from 9-45 where higher scores indicate a more positive attitude toward weight management.
Change in H-SCALE: Physical Exercise Score | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  The H-SCALE: Physical Exercise subscale is scored from 0-14 where higher scores indicate a more positive behavior toward physical exercise.
Change in H-SCALE: Smoking Exposure Score | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  The H-SCALE: Smoking Exposure subscale is scored from 0-14 where a score of 0 indicates a more positive attitude toward smoking exposure.
Change in H-SCALE: Alcohol Intake Score | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  The H-SCALE: Alcohol Intake subscale contains three questions and is scored as abstainer (does not drink) or non-adherent (reported drinking alcohol).
Change in H-SCALE: Healthy Eating Plan Score | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  The H-SCALE: Healthy Eating Plan subscale is scored from 0-70 where higher scores indicate a more positive attitude toward healthy eating.
Change in selected items from the Patient Assessment of Chronic Illness Care (PACIC) survey | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  PACIC will be scored on a likert scale from 1-5 (almost never to almost always) where higher scores indicate better assessment of chronic illness care.
Change in global hypertension care satisfaction score | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  Scored from 1-5 where higher scores indicate less satisfaction with hypertension care.
Change in pill count adherence ratio (PCAR) | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  PCAR is the total number of doses dispensed less that total doses missed divided by the total doses dispensed.
Change in self-reported adherence | Baseline, 6 months, 12 months (all participants assessed to 6 months, but participants on study early may also be assessed at 12, 18 and 24 months)
  Self-reported adherence is rated on a five point scale of how often patients are taking their medications as directed, from "less than half the time" to "100% of the time".
Proportion of lifestyle knowledge questions answered correctly | through study completion, an average of 12 months
  The proportion of a set of true-false or multiple choice questions developed for this study to assess hypertension-related lifestyle knowledge answered correctly

OTHER OUTCOMES:
Participant retention at 6 and 12 months | 6 months, 12 months
Proportion of possible study visits completed at 6 and 12 months | 6 months, 12 months
Mean duration of study visits | up to 24 months
Mean duration of physician review and care coordination time per patient encounter | up to 24 months
Comparison of antihypertensive medications prescribed and dosages | up to 24 months
Proportion of patients with an indication taking aspirin | up to 24 months
Proportion of patients taking two or more antihypertensives | up to 24 months
Estimated cost of care | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sean Duffy, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Community, San Lucas Tolimán, Guatemala

IPD SHARING:
Plan to Share IPD: No